CLINICAL TRIAL: NCT05558722
Title: Anlotinib Plus Chemotherapy as Neoadjuvant Treatment of High-risk, Early-stage Human Epidermal Growth Factor Receptor 2 (HER2)-Negative Breast Cancer: A Prospective, Single-arm, Single-center, Phase II Clinical Study
Brief Title: Anlotinib Combined With Chemotherapy and Neoadjuvant Therapy for Hormone Receptor-positive HER-2 Negative Breast Cancer
Acronym: ACNTBC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20202075-F-2
Record Dates: First submitted 2022-07-19; First posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Breast Cancer Stage II
Keywords: Breast cancer Antivascular drugs Neoadjuvant therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — anlotinib

STUDY DESIGN:
Intervention Model Description: Assigned to receive chemotherapy plus oral Anlotinib (12 mg qd, d1-14; 21 days per cycle; total 5 cycles)，chemotherapy comprised of pirarubicin at 50 mg/m2 and cyclophosphamide at 500 mg/m2 and albumin-bound paclitaxel at 200 mg/m2, (d1, 21 days per cycle; both total 6 cycles), which was then followed by surgery.
Masking Description: Check all roles that are masked or check None.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib (Experimental): Anlotinib is an oral multi-targeted tyrosine kinase inhibitor (TKI) that strongly inhibits VEGFR, PDGFR, FGFR, and c-kit. Anlotinib (12 mg qd, d1-14; 21 days per cycle; total 5 cycles) Combined TAC×6 cycles.
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: Anlotinib — Anlotinib (12 mg qd, d1-14; 21 days per cycle; total 5 cycles) Combined TAC×6 cycles: albumin-bound paclitaxel (200mg/m2, 1d Q3W) + pirarubicin （50mg/m2, 1d Q3W) + cyclophosphamide (500mg/m2, 1d Q3W);
  Other Names: TAC

SUMMARY:
Anlotinib is an oral multi-targeted tyrosine kinase inhibitor (TKI) that strongly inhibits VEGFR, PDGFR, FGFR, and c-kit. Combining anti-angiogenesis with chemotherapy yielded increased response rates in patients with early-stage human epidermal growth factor receptor 2 (HER2)-negative breast cancer. This study aims to evaluate the efficacy and safety of adding anlotinib to standard neoadjuvant chemotherapy in primary (HER2)-negative breast cancer. Patients aged 18 years or older with previously untreated stage ⅡB-IIIA histologically documented (HER2)-negative breast cancer were assigned to receive chemotherapy plus oral Anlotinib. The primary endpoint was pathologic complete response (pCR) (no invasive carcinoma in breast or axilla). Secondary end points included safety and disease-free survival (DFS).

DETAILED DESCRIPTION:
Anlotinib is an oral multi-targeted tyrosine kinase inhibitor (TKI) that strongly inhibits VEGFR, PDGFR, FGFR, and c-kit. Combining anti-angiogenesis with chemotherapy yielded increased response rates in patients with early-stage human epidermal growth factor receptor 2 (HER2)-negative breast cancer. This phase II study aims to evaluate the efficacy and safety of adding anlotinib to standard neoadjuvant chemotherapy in primary (HER2)-negative breast cancer.

Patients aged 18 years or older with previously untreated stage ⅡB-IIIA histologically documented (HER2)-negative breast cancer were assigned to receive chemotherapy plus oral Anlotinib (12 mg qd, d1-14; 21 days per cycle; total 5 cycles). Chemotherapy comprised of pirarubicin at 50 mg/m2 and cyclophosphamide at 500 mg/m2 and albumin-bound paclitaxel at 200 mg/m2, (d1, 21 days per cycle; both total 6 cycles), which was then followed by surgery. The primary endpoint was pathologic complete response (pCR) (no invasive carcinoma in breast or axilla). Secondary end points included safety and disease-free survival (DFS). Stratification was based on the clinical breast cancer stage .

ELIGIBILITY:
Inclusion Criteria:

* All patients were HER2 negative, deﬁ ned as munohistochemistry of 0/1+, or if 2+, ﬂ uorescence insitu hybridisation showed no evidence of ampliﬁ cation of the HER2 gene.
* Patients were required to have a palpable primary tumor at least 2.0 cm in diameter in the breast, as assessed by physical examination, and to be classified as having tumor stage T1c to T3, nodal stage N0 to N2a, and metastasis stage M0.
* Other eligibility criteria adequate cardiac function (left ventricular ejection fraction within the normal institutional range, as assessed by multiplegated acquisition scan or echocardiogram), adequate bone marrow, hepatic, and renal function, and appropriate Eastern Cooperative Oncology Group (ECOG) performance status (0-2).
* All patients provided written informed consent.

Exclusion Criteria:

* Previously received anti-angiogenesis targeted drug therapy.
* patients have previous diagnosis of ischaemic heart disease, cerebrovascular disease, peripheral vascular disease, arterial or venous thromboembolic disease, cardiac failure, gastroduodenal ulcer, symptomatic diverticulitis, or inflammatory bowel disease.
* Previously received chemotherapy, radiotherapy, or endocrine therapy as treatment for breast cancer was allowed.
* No uncont rolled hypertension.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-30 (Estimated); Primary Completion 2023-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
pCR( pathological complete remission) | 8 weeks
  Pathological complete remission rate assessed by the investigator

SECONDARY OUTCOMES:
ADR | 8 weeks
  Adverse Drug Reactions
DFS | 8 weeks
  DFS(Disease-free survival)

CONTACTS AND LOCATIONS:
Overall Officials: Ting Wang, PhD, Principal Investigator — Xijing Hospital Affiliated to Air Force Military Medical University
Locations (1):
- Xijing Hospital Affiliated to Air Force Military Medical University, Xi'an, Shannxi Province, China

IPD SHARING:
Plan to Share IPD: Undecided